CLINICAL TRIAL: NCT07107230
Title: A Phase 1 Study of JNJ-95437446 in Participants With Advanced-Stage Solid Tumors
Brief Title: A Study of JNJ-95437446 in Participants With Advanced-Stage Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 95437446LUC1001; 95437446LUC1001 (Other: Janssen Research & Development, LLC); 2025-521535-36-00 (Registry Identifier: EUCT number)
Record Dates: First submitted 2025-08-05; First posted 2025-08-06 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Colorectal Neoplasms
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- JNJ-95437446 (Experimental): Participants will receive JNJ-95437446 in Part 1 until at least two recommended phase 2 doses (RP2Ds) has been developed. Participants in Part 2 will receive JNJ-95437446 at the RP2Ds developed in Part 1.
  Interventions: Drug: JNJ-95437446

INTERVENTIONS:
Drug: JNJ-95437446 — JNJ-95437446 will be administered.

SUMMARY:
The purpose of this study is to determine recommended phase 2 doses (RP2Ds) of JNJ-95437446 in Part 1, and to further evaluate the safety of the RP2Ds in participants with advanced solid tumors in Part 2.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have been previously diagnosed with histologically confirmed unresectable, locally advanced, or metastatic non-small cell lung cancer, colorectal carcinoma, or head and neck squamous cell carcinoma
* Participants with non-small cell lung cancer (NSCLC) adenocarcinoma and colorectal cancer (CRC) must have local molecular testing to determine epidermal growth factor receptor (EGFR) mutational status for NSCLC and Kirsten rat sarcoma/neuroblastoma ras viral oncogene/v-raf murine sarcoma oncogene B1 (KRAS/NRAS/BRAF) mutation status for CRC
* Have measurable or evaluable disease:
* Part 1: Either measurable or evaluable disease; Part 2: At least 1 measurable lesion per response evaluation criteria in solid tumors (RECIST) version (v) 1.1
* Have an eastern cooperative oncology group (ECOG) performance status of 0 to 1 at screening
* Participants must have appropriate hematologic, renal, and hepatic function within the required limits

Exclusion Criteria:

* Any prior medical history of ILD/pneumonitis, including pneumonitis from anti-PD-1/ PD-L1 antibody or radiation that required systemic steroids
* Toxicity from prior anticancer therapy that has not resolved to Grade <=1
* Evidence of clinically significant active viral, bacterial, or fungal infection within 7 days before the first dose of study treatment requiring systemic or non-topical treatment
* History of clinically significant cardiovascular disease within 6 months prior to signing informed consent
* Participants with prior or concurrent second malignancy cannot be enrolled if prior/concurrent malignancy's natural history of treatment is likely to interfere with any safety or efficacy study endpoints

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 380 (Estimated)
Dates: Start 2025-07-15 (Actual); Primary Completion 2027-11-18 (Estimated); Study Completion 2028-04-24 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events (AEs) by Severity | Up to 2 years and 4 months
  An AE is any untoward medical occurrence in a clinical study participant administered a pharmaceutical (investigational or non-investigational) product and does not necessarily have a causal relationship with the intervention. Severity will be graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 5.0. Severity scale ranges from Grade 1 (Mild) to Grade 5 (Death). Grade 1= Mild, Grade 2= Moderate, Grade 3= Severe, Grade 4= Life-threatening and Grade 5= Death related to adverse event.
Part 1: Number of Participants with Dose-Limiting Toxicity (DLT) | Up to 21 days
  The DLTs are specific adverse events that includes high grade hematologic or non-hematologic toxicities with exceptions and/or toxicities leading to treatment discontinuation.

SECONDARY OUTCOMES:
Objective Response Rate | Up to 2 years and 4 months
  Objective response rate (ORR) is defined as the percentage of participants who have best response of complete response (CR) or partial response (PR) according to response evaluation criteria in solid tumors (RECIST).
Duration of Response (DOR) | Up to 2 years and 4 months
  DOR is defined for the responders from the date of initial documentation of a response to the date of first documented evidence of disease progression according to RECIST version (v.) 1.1, or death due to any cause, whichever occurs first.
Progression Free Survival (PFS) | Up to 2 years and 4 months
  PFS is defined as the time from the first dose of JNJ-95437446 to either progressive disease (PD) or death due to any cause, whichever comes first.
Maximum Plasma Concentration (Cmax) for JNJ-95437446 | Up to 2 years and 4 months
  Serum samples will be analyzed to determine Cmax of JNJ-95437446 antibody-drug conjugate, total antibody, released payload and the payload's metabolite.
Time to Reach Cmax (Tmax) for JNJ-95437446 | Up to 2 years and 4 months
  Tmax defined as the the time to reach maximum observed plasma concentration of JNJ-95437446 antibody-drug conjugate, total antibody, released payload and the payload's metabolite will be reported.
Area Under the Plasma Concentration - Time (AUC [0-t]) Curve for JNJ-95437446 antibody-drug conjugate, total antibody, released payload and the payload's metabolite. | Up to 2 years and 4 months
  AUC (0-t) defined as area under the plasma concentration-time curve during a dosing interval of JNJ-95437446 antibody-drug conjugate, total antibody, released payload and the payload's metabolite will be reported.
Number of Participants With Anti JNJ-95437446 Antibodies | Up to 2 years and 4 months
  Serum samples will be analyzed for the detection of anti-JNJ-95437446 antibodies using a validated assay method.

CONTACTS AND LOCATIONS:
Locations (6):
- United States (2):
  - Florida Cancer Specialists, Sarasota, Florida
  - NEXT Oncology, Fairfax, Virginia
- South Korea (2):
  - Severance Hospital Yonsei University Health System, Seoul
  - Samsung Medical Center, Seoul
- Spain (2):
  - Hosp. Univ. 12 de Octubre, Madrid
  - Hosp Univ Hm Sanchinarro, Madrid

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of Johnson & Johnson Innovative Medicine is available at innovativemedicine.jnj.com/our-innovation/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://innovativemedicine.jnj.com/our-innovation/clinical-trials/transparency